CLINICAL TRIAL: NCT04726527
Title: Clinical Evaluation of Florbetapir F 18 (18F-AV-45) / Determinants of Neurodegenerative Decline in Primary Progressive Aphasia
Brief Title: Clinical Evaluation of Florbetapir in Primary Progressive Aphasia
Acronym: PPA
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB23-1391
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Primary Progressive Aphasia; Alzheimer Disease; Dementia
Keywords: Alzheimer's Disease; Dementia; Primary Progressive Aphasia; Neurocognitive Disorders; Speech Disorders
MeSH Terms: conditions — Aphasia, Primary Progressive; Alzheimer Disease; Dementia; Neurocognitive Disorders; Speech Disorders | interventions — florbetapir; Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Florbetapir F 18 Recipients: Participants in this arm of the study will receive a 10 mCi (370 MBq) bolus injection of florbetapir F 18 and then be scanned in a PET scanner for brain imaging.
  Interventions: Drug: Florbetapir F 18; Device: Positron Emission Tomography

INTERVENTIONS:
Drug: Florbetapir F 18 — A single injection of 10 mCi (370 MBq) florbetapir F 18 will be administered by intravenous bolus injection.
  Other Names: trade name Amyvid
Device: Positron Emission Tomography — PET Scan for brain imaging
  Other Names: PET

SUMMARY:
The purpose of this research is to better understand how dementia affects activity in different parts of the brain.

DETAILED DESCRIPTION:
This study is being done to examine the usefulness of Positron Emission Tomography (PET) imaging with florbetapir F 18 as a biomarker in the identification of amyloid-ß peptide (Aß) in the brain. Amyloid-ß peptide (Aß) accumulates in the brains of patients with Alzheimer's disease. Florbetapir F 18 sticks to the amyloid plaques in the brain and emits a low level of gamma rays which can be detected by a PET camera. The development of biomarker and imaging studies that track the development of PPA and reflect the change in people's bodies may help other people who have a similar medical problem in the future.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can tolerate the PET scan procedures

Exclusion Criteria:

* Clinically significant cardiovascular disease
* clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances
* Pregnant
* Breastfeeding
* Women of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception.
* History of relevant severe drug allergy or hypersensitivity
* Patients who have received an investigational medication under an FDA Investigational New Drug (IND) protocol within the last 30 days.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from other research projects at Northwestern's Mesulam Center. Some of these projects recruit participants from the local Chicagoland area and others recruit participants from across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2015-09-02 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Detecting amyloid burden in subjects with neurodegenerative diseases | 4 years
  The study will provide standardized conditions for florbetapir F 18 use, amyloid binding as measured by PET imaging, and long-term outcome in cognitively normal volunteers, patients with Alzheimer's Disease, patients with Mild Cognitive Impairment, and patients with other neurodegenerative diseases. It will also facilitate evaluation of subject's amyloid burden in companion studies such as longitudinal studies of aging, studies of progressive cognitive impairment, and studies of imaging and blood/cerebrospinal fluid biomarkers of neurodegenerative disease.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rogalski, Ph.D, Principal Investigator — University of Chicago
Locations (1):
- The Healthy Aging & Alzheimer's Research Care Center - University of Chicago, Chicago, Illinois, United States